CLINICAL TRIAL: NCT04623255
Title: A Randomised Controlled Trial of Plasma Exchange With Standard of Care Compared to Standard of Care Alone in the Treatment of Severe COVID-19 Infection (COVIPLEX)
Brief Title: Study of Plasma Exchange in Severe COVID-19
Acronym: COVIPLEX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132796
Record Dates: First submitted 2020-06-11; First posted 2020-11-10 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Plasma Exchange

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STANDARD OF CARE (No Intervention): Standard patient care for severe COVID-19
- Plasma exchange (Active Comparator): Standard patient care for severe COVID-19 with. plasma exchange daily for 5 days x 3 courses as required
  Interventions: Drug: OCTAPLAS

INTERVENTIONS:
Drug: OCTAPLAS — plasma exchange
  Other Names: plasma exchange
  Arms: Plasma exchange

SUMMARY:
The rationale in severe COVID19 infection is to undertake PEX to aid reduction of the hyperinflammation and reduce the morbidity and mortality to the lungs, but also systemically, such as the heart, kidneys and brain. A feasibility study of PEX therapy has been undertaken and confirmed a reduction in the inflammatory markers, no VTE/arterial events and normalisation of the renal function and cardiac function throughout the period of therapy. As plasma exchange is an intensive treatment modality, blocks of 5 daily PEX will be undertaken. Further blocks of PEX treatment can be initiated as dictated by the clinical and laboratory parameters. Unlike many therapeutic schedules, there is no immunosuppression associated with PEX; indeed, the resulting decrease in inflammatory markers were shown to be associated with an increase and sustained lymphocytes count.

DETAILED DESCRIPTION:
COVID19 is a viral pandemic associated with primarily respiratory pathology, in the form of microvascular and macrovascular thrombosis. In patients requiring hospital admission, there is severe disease, requiring respiratory support, from high dose oxygen therapy or ventilatory assistance, which may be invasive or non invasive. The pathology of COVID19 is poorly understood, but it is accepted there is an inflammatory-thrombotic basis. Despite current therapeutic platforms, there is no consensus on a specific therapy within a trial setting that has proven benefit in severe COVID 19.

Thrombotic microangiopathies, such as TTP, are a different disease, but have a comparable prothrombotic phenotype, and similar or higher inflammatory parameters, including D Dimers, ferritin, LDH and IL-6 at acute presentation and resolve with plasma exchange (PEX). The rationale in severe COVID19 infection is to undertake PEX to aid reduction of the hyperinflammation and reduce the morbidity and mortality to the lungs, but also systemically, such as the heart, kidneys and brain. A feasibility study of PEX therapy has been undertaken and confirmed a reduction in the inflammatory markers, no VTE/arterial events and normalisation of the renal function and cardiac function throughout the period of therapy. As plasma exchange is an intensive treatment modality, blocks of 5 daily PEX will be undertaken. Further blocks of PEX treatment can be initiated as dictated by the clinical and laboratory parameters. Unlike many therapeutic schedules, there is no immunosuppression associated with PEX; indeed, the resulting decrease in inflammatory markers were shown to be associated with an increase and sustained lymphocytes count. Therefore, as patients with COVID-19 have elevated procoagulant factors including VWF and factor VIII secondary to direct endothelial activation. This is associated with an exaggerated pro-inflammatory immune response and microvascular thrombosis; resulting in multi-organ dysfunction and eventually death. PEX will improve coagulopathy, as measured by VWF:ADAMTS 13 ratio and D Dimers, with an associated reduction in inflammation, organ-related microthrombosis, and ventilatory support.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Proven COVID-19/high clinical suspicion of COVID-19
* Hypoxia/respiratory compromise defined as requiring respiratory support of >2L/min of oxygen by nasal cannulae to maintain SpO2<96%.
* Raised inflammatory parameters: at least 2 of the following:

  1. Raised LDH (> 2 x ULN)
  2. Raised D Dimers (> 2X ULN)
  3. Raised CRP (>2X ULN)
* Females of childbearing potential have a negative pregnancy test within 7 days prior to being randomised. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal

Exclusion Criteria:

* Significant co-morbid illness with treatment escalation limited to CPAP

  * Active bleeding
  * PF ratio < 100 on mechanical ventilation OR noradrenaline requirement > 0.5mcg/kg/min to maintain MAP > 65mmHg (suggests futility)
  * Known allergies to Octaplas or excipients
  * Females who are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Scully, MD, Principal Investigator — UCLH
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arulkumaran N, Thomas M, Stubbs M, Prasanna N, Subhan M, Singh D, Ambler G, Waller A, Singer M, Brealey D, Scully M. A randomised controlled trial of plasma exchange compared to standard of care in the treatment of severe COVID-19 infection (COVIPLEX). Sci Rep. 2024 Jul 23;14(1):16876. doi: 10.1038/s41598-024-67028-3. PMID 39043682

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | STANDARD OF CARE | Plasma Exchange
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Note: 23 patients with severe COVID-19 were randomised. One patient withdrew from the study 1 day after randomisation and their data has been excluded from the analysis. 11 were randomised to the treatment group receiving at least one course of Plasma Exchange (PEX).11 were assigned to the control group receiving only standard of care treatment (SOC). There were no follow-up data for a further two participants (1 from each arm) and hence they were omitted from this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | STANDARD OF CARE | Plasma Exchange | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 9 | 10 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7 | 4 | 11
  Asian | 1 | 4 | 5
  Black | 2 | 2 | 4
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Inflammatory Marker Reduction of at Least 50% at Any Efficacy Time Point
Description: The primary outcome in this study is a binary outcome indicating whether there was a reduction of at least 50% (compared to baseline) in two or more inflammatory markers [CRP, LDH, D-Dimer] during a"comparable duration of treatment" with either PEX or Standard of Care after study initiation.
Time Frame: The inflammatory markers recorded in this study are C reactive protein (CRP), lactate dehydrogenase(LDH) and D-Dimer, and we consider whether there is a reduction during the designated follow-up period (i.e. follow-up days 6, 7, 14, 21 and 28).
Population: Note: 23 patients with severe COVID-19 were randomised. One patient withdrew from the study 1 day after randomisation and their data has been excluded from the analysis. There were no follow-up data for a further two participants for this endpoint (1 from each arm) and hence they were omitted from this analysis, so data from a total of 20 participants was analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | STANDARD OF CARE | Plasma Exchange
Number analyzed (Participants) | 10 | 10
Participants | 5 | 8
Statistical Analysis 1: Comparison: STANDARD OF CARE vs Plasma Exchange; The primary analysis will involve a comparison of the binary outcome '50% reduction in at least two inflammation markers' between the PEX and Standard of Care (control) trial arms using a chi-squared test. The risk difference (and ratio) will be estimated with a 95% confidence interval; Test type: Superiority; p = 0.16, Chi-squared

2. Primary Outcome: Change in Inflammatory Marker-CRP
Description: To compare the change in inflammatory marker CRP with Plasma Exchange and control groups in patients with severe COVID-19.
  Measured as number of participants who experienced a reduction of 50% at any follow-up time point.
Time Frame: We consider whether there is a reduction in inflammatory marker CRP during the designated follow-up period (i.e. follow-up days 6, 7, 14, 21 and 28).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STANDARD OF CARE | Plasma Exchange
Number analyzed (Participants) | 10 | 10
Participants | 8 | 7
Statistical Analysis 1: Comparison: STANDARD OF CARE vs Plasma Exchange; The primary analysis will involve a comparison of the binary outcome '50% reduction in inflammation marker CRP' between the PEX and Standard of Care (control) trial arms using a chi-squared test. The risk difference (and ratio) will be estimated with a 95% confidence interval; Test type: Superiority; p = 0.606, Chi-squared

3. Primary Outcome: Change in Inflammatory Marker-D Dimer
Description: To compare the change in inflammatory marker D-dimer with Plasma Exchange and control groups in patients with severe COVID-19.
  Measured as number of participants who experienced a reduction of 50% at any follow-up time point.
Time Frame: We consider whether there is a reduction in inflammatory marker D-dimer during the designated follow-up period (i.e. follow-up days 6, 7, 14, 21 and 28).
Population: Note: 23 patients with severe COVID-19 were randomised. One patient withdrew from the study 1 day after randomisation and their data has been excluded from the analysis. There were no follow-up data for a further three participants for this endpoint (1 from standard of care arm and 2 from plasma exchange arm) and hence they were omitted from this analysis, so data from a total of 19 participants was analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | STANDARD OF CARE | Plasma Exchange
Number analyzed (Participants) | 10 | 9
Participants | 4 | 6
Statistical Analysis 1: Comparison: STANDARD OF CARE vs Plasma Exchange; The primary analysis will involve a comparison of the binary outcome '50% reduction in inflammation marker D-Dimer' between the PEX and Standard of Care (control) trial arms using a chi-squared test. The risk difference (and ratio) will be estimated with a 95% confidence interval; Test type: Superiority; p = 0.245, Chi-squared

4. Primary Outcome: Change in Inflammatory Marker-LDH
Description: To compare the change in inflammatory marker LDH with Plasma Exchange and control groups in patients with severe COVID-19.
  Measured as number of participants who experienced a reduction of 50% at any follow-up time point.
Time Frame: We consider whether there is a reduction in inflammatory marker LDH during the designated follow-up period (i.e. follow-up days 6, 7, 14, 21 and 28).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | STANDARD OF CARE | Plasma Exchange
Number analyzed (Participants) | 10 | 10
Participants | 5 | 6
Statistical Analysis 1: Comparison: STANDARD OF CARE vs Plasma Exchange; The primary analysis will involve a comparison of the binary outcome '50% reduction in inflammation marker LDH' between the PEX and Standard of Care (control) trial arms using a chi-squared test. The risk difference (and ratio) will be estimated with a 95% confidence interval; Test type: Superiority; p = 0.653, Chi-squared

ADVERSE EVENTS:
Time Frame: All adverse events will be recorded from consent to the end of trial (day 28 after randomisation).
Description: Serious Adverse Events associated with COVID-19 infection were not reported to Sponsor for this trial, however they were recorded in the database and are included in this report.
Arm/Group | STANDARD OF CARE | Plasma Exchange
All-Cause Mortality (participants affected / at risk) | 1/11 | 2/11
Serious Adverse Events (participants affected / at risk) | 4/11 | 6/11
Other Adverse Events (participants affected / at risk) | 11/11 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STANDARD OF CARE (N=11) | Plasma Exchange (N=11)
Blood pressure decreased (Investigations) | 0 (0) | 1 (2)
Body temperature increased (Investigations) | 1 (1) | 1 (1)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 2 (5)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Oxygen therapy (Surgical and medical procedures) | 1 (1) | 2 (2)
Drug therapy (Surgical and medical procedures) | 1 (1) | 0 (0)
Endotracheal intubation (Surgical and medical procedures) | 2 (2) | 4 (4)
Lung assist device therapy (Surgical and medical procedures) | 1 (1) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Central nervous system infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STANDARD OF CARE (N=11) | Plasma Exchange (N=11)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (2) | 0 (0)
Oxygen therapy (Surgical and medical procedures) | 2 (2) | 0 (0)
Intensive care (Surgical and medical procedures) | 1 (1) | 0 (0)
Endotracheal intubation complication (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Wound secretion (General disorders) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 2 (2) | 1 (2)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Body temperature abnormal (Investigations) | 1 (1) | 1 (4)
Body temperature increased (Investigations) | 1 (1) | 1 (1)
Coma scale abnormal (Investigations) | 1 (1) | 0 (0)
Computerised tomogram thorax (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Drug monitoring procedure incorrectly performed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth loss (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (4)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Tracheostomy (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT04623255/Prot_SAP_000.pdf